CLINICAL TRIAL: NCT00072332
Title: A Phase I Dose Escalation Study of Edotecarin (PHA-782615) and Cisplatin in Adult Patients With Advanced/Metastatic Solid Tumors
Brief Title: Edotecarin and Cisplatin in Treating Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000339607; MSKCC-03070; PHARMACIA-EDOAES-2730-001
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2009-12

CONDITIONS: Esophageal Cancer; Gastric Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; stage IV esophageal cancer; stage IV gastric cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Cisplatin; edotecarin

INTERVENTIONS:
Drug: cisplatin
Drug: edotecarin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as edotecarin and cisplatin, use different ways to stop tumor cells from dividing so they stop growing or die. Combining edotecarin with cisplatin may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining edotecarin with cisplatin in treating patients who have advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and recommended phase II dose of edotecarin when administered with cisplatin (administered in 2 different schedules) in patients with advanced or metastatic solid tumors.

Secondary

* Determine the safety profile of this regimen in these patients.
* Determine the plasma pharmacokinetics of this regimen in these patients.
* Determine the antitumor activity of this regimen in these patients.

OUTLINE: This is an open-label, multicenter, dose-escalation study of edotecarin. Patients are assigned to 1 of 2 schedules.

* Schedule A: Patients receive cisplatin IV over 30 minutes and edotecarin IV over 1 hour on days 1 and 8.
* Schedule B: Patients receive cisplatin IV over 2 hours and edotecarin IV over 1 hour on day 1.

In both schedules, courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients in each schedule receive escalating doses of edotecarin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 10 additional patients with metastatic esophageal or gastric cancer receive treatment as above at the MTD.

Patients are followed every 2 months for 1 year or until disease progression.

PROJECTED ACCRUAL: A maximum of 80 patients (40 per schedule) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Histologically or cytologically confirmed active solid tumor malignancy
  * Histologically confirmed esophageal or gastric cancer* meeting all the following criteria:

    * Previously untreated disease
    * Metastatic disease
    * Measurable disease

      * At least 1 unidimensionally measurable lesion at least 20 mm by conventional techniques OR 10 mm by spiral CT scan NOTE: *Patients with esophageal or gastric cancer are enrolled after the maximum tolerated dose has been determined
* No known brain or leptomeningeal disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN) (regardless of liver involvement by tumor)
* SGOT no greater than 3 times ULN (5 times ULN if there is liver involvement by tumor)
* Albumin at least 3.0 g/dL

Renal

* Creatinine no greater than 1.5 mg/dL

Cardiovascular

* None of the following within the past 12 months:

  * Myocardial infarction
  * Severe/unstable angina
  * Symptomatic congestive heart failure
  * Cerebrovascular accident
  * Transient ischemic attack
  * Deep vein thrombosis
  * Other significant thromboembolic event
* No ongoing grade 2 or greater cardiac dysrhythmia
* No atrial fibrillation

Pulmonary

* No pulmonary embolism within the past 12 months

Gastrointestinal

* No active inflammatory bowel disease
* No partial or complete bowel obstruction
* No chronic diarrhea

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No grade 2 or greater acute toxic effects
* No active infection
* No other concurrent acute or chronic medical or psychiatric condition or laboratory abnormality that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior treatment with any of the following systemic therapies for metastatic cancer*:

  * Antibody therapy
  * Immunotherapy
  * Gene therapy
  * Vaccine therapy
  * Cytokine therapy
  * Inhibitors of vascular endothelial growth factor/Flk-1 pathway
* No concurrent sargramostim (GM-CSF)
* No concurrent antibody therapy or immunotherapy NOTE: *Patients with esophageal or gastric cancer only

Chemotherapy

* No more than 1 prior chemotherapy regimen for metastatic disease*
* No prior high-dose chemotherapy requiring hematopoietic stem cell rescue
* No other concurrent chemotherapy NOTE: *No prior chemotherapy for metastatic disease for patients with esophageal or gastric cancer

Endocrine therapy

* No concurrent hormonal treatment

Radiotherapy

* No prior radiotherapy to more than 25% of bone marrow reserve
* No prior radiotherapy to the sole measurable lesion*
* No concurrent radiotherapy NOTE: *Patients with esophageal or gastric cancer only

Surgery

* More than 12 months since prior coronary/peripheral artery bypass graft surgery

Other

* Recovered from prior therapy
* More than 6 months since last dose of prior adjuvant therapy*
* No prior treatment with any of the following systemic therapies for metastatic cancer*:

  * Cyclooxygenase-2 inhibitors
  * Matrix metalloprotease inhibitors
  * Epidermal growth factor receptor inhibitors
  * Other experimental agents
* No other concurrent anticancer therapy
* No concurrent enrollment in another clinical trial
* No other concurrent experimental drugs NOTE: *Patients with esophageal or gastric cancer only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08; Primary Completion 2005-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Ilson, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States